CLINICAL TRIAL: NCT02438046
Title: Platelet Rich Fibrin in the Treatment of Palatal Wounds After Epithelialized Free Gingival Grafts Harvesting. A Randomized Clinical Trial
Brief Title: Platelet Rich Fibrin in the Treatment of Palatal Wounds
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Michele Paolantonio, Full time professor, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1/2015
Record Dates: First submitted 2015-04-27; First posted 2015-05-08 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Gingival Recession
Keywords: Connective Tissue Grafts; Wound healing; Biomaterials; Pain; Clinical Trials; Mucogingival Surgery
MeSH Terms: conditions — Gingival Recession; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palatal wound bandage by PRF (Experimental): Intervention: In the test group (n=20 patients) the palatal wound will be protected by a quadruple layer of Platelet Rich Fibrin obtained by folding on itself 2 Platelet Rich Fibrin membranes
  Interventions: Procedure: Palatal wound bandage
- Palatal wound bandage by gelatin sponge (Placebo Comparator): Intervention: The control group patients (n=20) will have their palatal wound medicated by absorbable gelatin sponge.
  Interventions: Procedure: Palatal wound bandage

INTERVENTIONS:
Procedure: Palatal wound bandage — Treatment of Palatal wounds by Platelet Rich Fibrin or absorbable gelatin sponge.

SUMMARY:
In this study it will be investigated the usefulness of Platelet-Rich Fibrin (PRF) on in the epithelialized connective tissue graft palatal donor site healing acceleration and in the patient's morbidity reduction. Forty patients, with at least one gingival recession will be treated by a coronally advanced flap (CAF) with connective tissue graft(CTG) resulting from the de-epithelialization of a free gingival graft. In the test group (20 patients) a quadruple layer of PRF membrane will be placed over the palatal wounds; conversely, the control group patients will be treated by an absorbable gelatin sponge. Patients will be monitored at 1, 2, 3 and 4 weeks after surgery for the complete re-epithelialization of the palatal wound (CWE), the alteration of sensibility (AS) around the wound area, the post-operative discomfort (D), and the changes of feeding habits (CFH) by a visual analogic scale (VAS) evaluation. Furthermore, the analgesics consumption and the existence of delayed bleeding from the palatal wound (DWB) during the first post-operative week will be assessed.

ELIGIBILITY:
Inclusion Criteria: are as follows:

* to have a single gingival recession to be treated by a mucogingival surgery intervention
* to be in good systemic health
* to have a good oral hygiene

Exclusion Criteria:

* no systemic diseases; no coagulation disorders; no medications affecting periodontal status in the previous 6 months; no pregnancy or lactation;
* no smoking habits;
* no periodontal surgery on the experimental sites;
* no inadequate endodontic treatment
* no tooth mobility at the site of surgery

Max Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is to assess the time needed to obtain a complete re epithelialization of the palatal wound | four weeks

CONTACTS AND LOCATIONS:
Locations (1):
- G. d'Annunzio University, Chieti, CH, Italy